CLINICAL TRIAL: NCT01312038
Title: A Pilot Study of the Effect of Simethicone in Adult Subjects With a Common Cold on Eustachian Tube Dysfunction
Brief Title: Effect of Simethicone on Eustachian Tube Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, William J. Doyle, Professor of Otolaryngology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO011010385
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Otitis Media
Keywords: Eustachian tube; otitis; middle-ear pressure; simethicone
MeSH Terms: conditions — Otitis Media; Otitis | interventions — Simethicone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- simethicone (Experimental): 125 mg tablet
  Interventions: Drug: Simethicone
- placebo (Placebo Comparator): chewable calcium tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simethicone — single 125 mg chewable tablet
  Arms: simethicone
Drug: Placebo — chewable calcium tablet
  Arms: placebo

SUMMARY:
This study is designed to measure the effects of a chewable Simethicone tablet taken by mouth on middle-ear pressure in adults with a common cold and evidence of abnormal middle-ear pressure. In children and adults, middle-ear diseases such as otitis media (the buildup of fluid within the middle ear) and a form of temporary hearing loss occur if the Eustachian tube does not open, does not open often enough or is always open. Simethicone, available over-the-counter under several brand names including Gas-X, may help break up the bubbles that may block the opening of the Eustachian tube in the back of the nose during a cold, allowing air to pass between the nose and middle ear. This study requires a single visit to the Middle Ear Physiology Laboratory in the Oakland section of Pittsburgh. If eligible for the study, Eustachian tube function testing will be done; the Simethicone tablet or placebo (a tablet that looks and tastes like the Simethicone tablet but has no active ingredient) will be given and Eustachian tube function testing repeated.

DETAILED DESCRIPTION:
For the Eustachian tube function testing, the subject and a technician are seated comfortably within a pressure chamber, a room-like chamber in which the air pressure can be varied much like in an airplane or submarine. Middle ear pressure will be measured in each ear by tympanometry, a test done by inserting a small probe (an earplug attached to a rubber or plastic tube that measures ear pressure) half-way into the ear canal and changing the pressure in the probe. Then, microphones will be placed in the ear canals and a sound source placed into one nostril. The chamber pressure is then decreased and increased to various pressures and middle ear pressure is measured at these various pressures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years
* Healthy subjects other than current upper respiratory tract infection ("cold")
* Jackson Score of 6 on screening
* Subject reports symptom onset within 4 days of entry visit
* Unilateral or bilateral middle-ear pressure <-50 mmH2O

Exclusion Criteria:

* Otoscopic diagnosis of unilateral or bilateral otitis media
* Presence of tympanostomy tubes or tympanic membrane perforations bilaterally
* Asthma or any chronic medical disease or condition
* Use of an "over the counter" medicine within 24 hours of study or prescription within 4 weeks of the study day (except birth control)
* Use of an experimental drug within 3 months of study
* An unusual or allergic reaction to simethicone, food dyes, or preservatives
* Pregnancy or breast feeding
* Ear surgery other than tympanostomy tube insertion

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Doyle, PhD, Principal Investigator — Department of Otolaryngology, Children's Hospital of Pittsburgh of UPMC
Locations (1):
- Middle Ear Physiology Laboratory of Children's Hospital of PIttsburgh of UPMC, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in March 2011 and was terminated in March 2013. Recruitment was done by advertisement in the community.
Pre-assignment Details: Ninety subjects (31 males, 59 females)were screened; 25 subjects entered the randomization phase.
Period: Overall Study
Arm/Group | Simethicone | Placebo
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis done by ears with evaluable tests.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simethicone | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (9.1) | 32.8 (11.7) | 29.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Fraction of Middle Ear (ME) Pressure Equilibrated (FGE)
Description: The proportion of the pressure chamber-ME pressure gradient equilibrated with 1 swallow
Time Frame: After achieving the desired ME-pressure chamber gradient at baseline and 30 min post treatment
Population: ears pre-treatment/ears post-treatment
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: ears
Groups:
- Simethicone-treated; Placebo: Outcome measure in each evaluable ear.
Arm/Group | Simethicone-treated | Placebo
Number analyzed (Participants) | 13 | 12
Number analyzed (ears) | 22 | 18
ratio
  Pre treatment FGE at -200 daPa | 0.17 (0.28) | 0.24 (0.34)
  post-treatment FGE at -200 daPa | 0.19 (0.28) | 0.23 (0.32)
  Pre -treatment FGE at 200 daPa | 0.24 (0.31) | 0.30 (0.34)
  Post-treatment FGE at 200 daPa | 0.24 (0.29) | 0.34 (0.37)
Statistical Analysis 1: Comparison: Simethicone-treated vs Placebo; Comparison of the simethicone and placebo groups with respect to the difference between the pre-post treatment FGE at ME-pressure chamber gradient of -200 daPa; Test type: Superiority or Other; p = 0.93, Paired T-test; df=34
Statistical Analysis 2: Comparison: Simethicone-treated vs Placebo; Comparison of the simethicone and placebo groups with respect to the difference between the pre-post treatment FGE at ME-pressure chamber gradient of 200 daPa; Test type: Superiority or Other; p = 0.39, Paired T-test; df = 31

ADVERSE EVENTS:
Time Frame: The subjects were assessed throughout the experimental procedure which lasted for 2 hours.
Arm/Group | Simethicone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No